CLINICAL TRIAL: NCT01839058
Title: Is Non-Cardiac Chest Pain Caused by Sustained Longitudinal Smooth Muscle Contraction?
Status: Completed | Type: Observational
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. William Paterson, Professor of Medicine, Queen's University
Other Study IDs: DMED-1559-13
Record Dates: First submitted 2013-04-16; First posted 2013-04-24 (Estimated); Results first posted 2017-08-03 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Chest Pain Atypical Syndrome
Keywords: Non Cardiac Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non Cardiac Chest Pain Patients: Patients with Chest Pain where Coronary Artery Disease has been formally ruled out are to undergo esophageal manometry testing.
  Interventions: Other: Esophageal Manometry
- Healthy Controls: Healthy volunteers without esophageal symptoms are to undergo esophageal manometry testing.
  Interventions: Other: Esophageal Manometry

INTERVENTIONS:
Other: Esophageal Manometry — Both cohorts will undergo standard high resolution esophageal manometry testing. This entails a catheter passed through the nose into the esophagus and measures pressure changes with a series of wet swallows. As part of the study, we will also be instilling both weak acid and saline into the esophagus.

SUMMARY:
Non-cardiac chest pain (NCCP) is a common disorder whose pathophysiology is poorly understood. Some evidence suggests it may be related to sustained esophageal contractions (SECs) of longitudinal smooth muscle. The investigators have previously shown that acid is a trigger for SECs and results in shortening of the esophagus. In this study, the investigators plan to prospectively evaluate esophageal shortening responses to acid in a group of patients with NCCP compared to controls. The investigators will use high resolution esophageal manometry coupled with acid infusion to evaluate shortening. The investigators hypothesize that at least a subset of patients with NCCP will have an exaggerated esophageal shortening response to acid which correlates with symptom production. If our hypothesis proves true, this may lead to a future therapeutic target in the treatment of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers:
* free of esophageal symptoms
* not on any acid suppressing medications
* Non Cardiac Chest Pain Patients:
* Angina like chest pain occuring at least once per month
* Coronary artery disease ruled out by stress test or angiogram

Exclusion Criteria:

* pre existing motility disorder of the esophagus
* connective tissue disease
* pregnancy
* taking calcium channel blockers, Nitrates, Gabapentin, Narcotics, Tricyclic antidepressants, Anti seizure medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with non cardiac chest pain as diagnosed by cardiologist or other physician. Healthy Volunteers will include anyone in the Kingston area who fulfils Inclusion and Exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Paterson, MD, FRCPC, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non Cardiac Chest Pain Patients | Healthy Controls
Started | 21 | 19
Completed | 17 | 16
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non Cardiac Chest Pain Patients | Healthy Controls | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (10.1) | 49.4 (18.3) | 50.9 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 7 | 9 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Esophageal Length With Acid
Description: Mean length of esophagus with acid infusion minus mean length of esophagus with saline infusion
Time Frame: Length at T= 20 minutes - Baseline (T=0)
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Non Cardiac Chest Pain Patients | Healthy Controls
Number analyzed (Participants) | 17 | 16
centimeters | -0.40 (0.54) | -0.39 (0.55)

2. Secondary Outcome: Esophageal Length at Symptom Onset
Description: Length of Esophagus as measured by manometry during acid infusion when patient reports symptoms
Time Frame: 20 minutes
Population: As pre-specified in the protocol, this Outcome Measure was intended to be analyzed only if a correlation was found between esophageal shortening and symptom production. Thus data was not collected.
Arm/Group | Non Cardiac Chest Pain Patients | Healthy Controls
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Esophageal Length at Maximal Symptom Intensity
Description: Mean length of esophagus at peak patient reported symptom intensity with acid infusion
Time Frame: 20 minutes
Population: Data Not collected given lack of correlation between symptoms and esophageal length.
Arm/Group | Non Cardiac Chest Pain Patients | Healthy Controls
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants for Whom a Correlation Was Found Between Symptom Onset and Esophageal Shortening
Description: Esophageal shortening will be defined as the point during the 20 minute acid infusion at which the lower esophageal sphincter begins to migrate proximally. A 2 minute window following this time point will then be used to determine if patients symptoms increased by > 2 on a visual analogue pain scale between 0 - 10.
Time Frame: 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Non Cardiac Chest Pain Patients | Healthy Controls
Number analyzed (Participants) | 17 | 16
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Non Cardiac Chest Pain Patients | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 0/21 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No